CLINICAL TRIAL: NCT01375491
Title: Blockade of Receptor Cleavage in Diabetes Mellitus With an MMP Inhibitor
Brief Title: Examination of the Anti-inflammatory and Insulin Sensitizing Properties of Doxycycline in Humans
Acronym: DOXY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Ruth L. Kirschstein National Research Service Award (U.S. Federal Agency); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 090395; 5M01RR000827 (NIH); P30DK063491 (NIH)
Record Dates: First submitted 2011-05-25; First posted 2011-06-17 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: doxycycline; insulin resistance; obesity; inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Insulin Resistance; Inflammation | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doxycycline (Experimental): Participants with DM2 receiving doxycycline 100mg BID
  Interventions: Drug: Doxycycline
- Placebo (Placebo Comparator): Pills prepared identical to doxycycline.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Doxycycline — generic doxycycline 100mg twice daily
  Other Names: Vibramycin
  Arms: Doxycycline
Other: Placebo — Placebo comparator to doxycycline
  Arms: Placebo

SUMMARY:
Obesity is a heightened state of inflammation in which production of cytokines and matrix metalloproteinases (MMPs) result in loss of function of insulin receptors and insulin resistance. Doxycycline (DOX) is a potent MMP inhibitor. We hypothesize that DOX will enhance insulin sensitivity and decreases inflammation in obese participants with type 2 diabetes (DM2).

DETAILED DESCRIPTION:
Design and Setting: 84 day (D84), double-blind, randomized, placebo (PL)-controlled clinical trial conducted in an academic tertiary care center.

Patients: Non-DM2 Controls (n=15); participants with DM2 receiving PL (n=13) or DOX (n=11).

Interventions: All participants were evaluated at day 1 (D1); those with DM2 were also evaluated at D84 after DOX 100mg twice daily or PL.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, medically stable, able to give informed consent, and comply with the protocol.
* Obesity with BMI >30 kg/m2.
* DM2 for less than 10 years.
* 7.5% < HA1C < 10%
* Taking insulin and/or oral medications (biguanide, sulfonlylurea, etc.)

Exclusion Criteria:

* Mental states that would preclude complete understanding of the protocol and compliance.
* Chronic illness such as renal failure (with creatinine clearance <80 ml/min for Specific Aim 2).
* Women of child-bearing age because of the potential hazard to the fetus (doxycycline may cause permanent discoloration of the teeth and deposition in bone inhibiting growth) and because doxycycline may render oral contraceptives less effective.
* Nursing mothers.
* Allergy to tetracyclines.
* Subjects taking the following drugs: penicillin or it's derivatives, anticoagulant therapy, antacids containing aluminum, calcium, or magnesium, iron-containing preparations, bismuth subsalicylate, barbiturates, carbamazepine, phenytoin or methoxyflurane, thiazolidinediones (TZD)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Herbst, PhD, MD, Principal Investigator — UCSD
Locations (1):
- University of California San Diego Clinical trials Research Institute, La Jolla, California, United States

REFERENCES:
- [Background] DeLano FA, Schmid-Schonbein GW. Proteinase activity and receptor cleavage: mechanism for insulin resistance in the spontaneously hypertensive rat. Hypertension. 2008 Aug;52(2):415-23. doi: 10.1161/HYPERTENSIONAHA.107.104356. Epub 2008 Jul 7. PMID 18606910
- [Result] Frankwich K, Tibble C, Torres-Gonzalez M, Bonner M, Lefkowitz R, Tyndall M, Schmid-Schonbein GW, Villarreal F, Heller M, Herbst K. Proof of Concept: Matrix metalloproteinase inhibitor decreases inflammation and improves muscle insulin sensitivity in people with type 2 diabetes. J Inflamm (Lond). 2012 Oct 1;9(1):35. doi: 10.1186/1476-9255-9-35. PMID 23025537

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study included non-type 2 diabetics controls (n = 15), and type two diabetics subjects randomized to placebo (n = 13) or doxycycline 100 mg twice daily (n = 11).
Groups:
- Doxycycline: Participants with DM2 receiving doxycycline 100mg BID
  Doxycycline : generic doxycycline 100mg twice daily
- Placebo: Pills prepared identical to doxycycline.
  Placebo : Placebo comparator to doxycycline
- Control: non- type two diabetics to serve as a control
Period: Overall Study
Arm/Group | Doxycycline | Placebo | Control
Started | 11 | 13 | 15
Completed | 9 | 12 | 15
Not Completed | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control: Participants enrolled without type 2 diabetes to serve as a control
- Total: Total of all reporting groups
Arm/Group | Doxycycline | Placebo | Control | Total
Number analyzed (Participants) | 11 | 13 | 15 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (1.9) | 54.5 (1.7) | 48.7 (3.1) | 54.9 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 5 | 9
  Male | 9 | 11 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: MMP Activity
Description: MMP activity is measured using a charge-changing peptide substrate for MMP-2 and MMP-9.
Time Frame: Baseline (Day 1)
Measure: Mean (Standard Error); unit: uM 5-FAM/h-ug protein
Groups:
- Control Arm: The study included non-DM2 controls (n = 15), but the non DM2 controls were not evaluated on day 84.
Arm/Group | Doxycycline | Placebo | Control Arm
Number analyzed (Participants) | 9 | 12 | 15
uM 5-FAM/h-ug protein | 56.8 (13.3) | 43.8 (4) | 47.2 (3.2)

2. Secondary Outcome: CRP
Description: Measure of global inflammation.
Time Frame: Baseline (Day 1)
Measure: Mean (Standard Error); unit: microgram/ml
Arm/Group | Doxycycline | Placebo | Control Arm
Number analyzed (Participants) | 9 | 11 | 15
microgram/ml | 7.4 (3.3) | 5.9 (1.8) | 1.9 (.8)
Statistical Analysis 1: Comparison: Doxycycline vs Placebo; See published paper; Test type: Superiority or Other; p < 0.05, ANOVA — See published paper; See published paper

3. Primary Outcome: MMP Activity
Description: MMP activity is measured using a charge-changing peptide substrate for MMP-2 and MMP-9. Only the Doxycycline and Placebo arms are reported because the control group was not evaluated at Day 84.
Time Frame: Day 84
Population: Only the Doxycycline and Placebo arms are reported because the control group was not evaluated at Day 84.
Measure: Mean (Standard Error); unit: uM 5-FAM/h-ug protein
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 9 | 12
uM 5-FAM/h-ug protein | 59.7 (4.3) | 56.6 (10.1)

4. Secondary Outcome: CRP
Description: Measure of global inflammation. Only the Doxycycline and Placebo arms are reported because the control group was not evaluated at Day 84.
Time Frame: Day 84
Population: Only the Doxycycline and Placebo arms are reported because the control group was not evaluated at Day 84.
Measure: Mean (Standard Error); unit: microgram/ml
Arm/Group | Doxycycline | Placebo
Number analyzed (Participants) | 9 | 11
microgram/ml | 2.3 (0.4) | 6.2 (1.8)

ADVERSE EVENTS:
Description: This information is being entered from a publication, since the Principal Investigator is no longer associated with the institution. The publication does not report on adverse events and so there is no way to report these numbers.
Arm/Group | Doxycycline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This information is being entered from a publication, since the Principal Investigator is no longer associated with the institution. The publication does not report on adverse events and so there is no way to report these numbers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No